Title of Study: Practices of Vitamin D Supplementation leading to Vitamin D toxicity:

**Experience from a Tertiary care center of a Low Middle Income Country** 

Manuscript type: Original article

**Date of Document:** 2<sup>nd</sup> November 2019

NCT Number: NCT05139576

## STATISTICAL ANALYSIS PLAN

The statistical analysis will be performed using the Microsoft Excel 2016. Subjects will be categorized into two age groups: <18 years (pediatric) and ≥18 years (adult). Frequencies of subjects with VD toxicity will be derived and their correlates will be evaluated in the both the age groups. Demographics (age and gender), calcium status of subjects, indications, formulation strengths, frequency, duration, cumulative and daily dose of supplementation will be generated. Descriptive statistics median (interquartile range, IQR) will be calculated for numerical data while frequency (percentage) for categorical data.

## **REFERENCES:**

- Khan AH, Igbal R, Naureen G, Dar FJ, Ahmed FN. Prevalence of vitamin D deficiency and its correlates: results of a community-based study conducted in Karachi, Pakistan. Arch Osteoporos.7(1-2):275-82.
- Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, et al. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011;96(7):1911-30.
- Dawson-Hughes B, Mithal A, Bonjour JP, Boonen S, Burckhardt P, Fuleihan GE, et al. IOF position statement: vitamin D recommendations for older adults. Osteoporos Int. 2010;21(7):1151-4.
- Deluca HF, Prahl JM, Plum LA. 1,25-Dihydroxyvitamin D is not responsible for toxicity caused by vitamin D or 25-hydroxyvitamin D. Arch Biochem Biophys. 505(2):226-30.

1

- 5. Taylor PN, Davies JS. A review of the growing risk of vitamin D toxicity from inappropriate practice. Br J Clin Pharmacol. 2018.
- 6. Shea RL, Berg JD. Self-administration of vitamin D supplements in the general public may be associated with high 25-hydroxyvitamin D concentrations. Ann Clin Biochem. 2017;54(3):355-61.
- 7. Khan AH, Majid H, Iqbal R. Shifting of vitamin D deficiency to hypervitaminosis and toxicity. J Coll Physicians Surg Pak. 2014;24(7):536.
- 8. Alshahrani F, Aljohani N. Vitamin D: deficiency, sufficiency and toxicity. Nutrients.5(9):3605-16.
- 9. Lowe H, Cusano NE, Binkley N, Blaner WS, Bilezikian JP. Vitamin D toxicity due to a commonly available "over the counter" remedy from the Dominican Republic. J Clin Endocrinol Metab.96(2):291-5.